CLINICAL TRIAL: NCT04596202
Title: The Effect of Position in Post-op Newborns Hospitalized in Pediatric Cardio Vascular Surgery Intensive Care Unit on Gastric Residual Volume and Comfort Level
Brief Title: The Effect of Position on Gastric Residual Volume and Comfort Level in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Fatma Yılmaz Kurt, Asist Prof Dr, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CanakkaleOMU
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Comfort; Newborn, Infant, Disease; Position; Residual
Keywords: Newborn; Comfort Score; Residual Volume; infant positioning
MeSH Terms: conditions — Disease | interventions — Supine Position; Prone Position

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Crossover Design Model
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supine Position (Experimental): It is the supine position. The body parts of the patient stand as if the patient is standing upright. The head, neck and shoulders should be supported with a pillow placed under the head. Arms are aside and body muscles are relaxed. The upper arms should lie on both sides of the body, should slightly be moved away from the body and should be supported by a pillow.
  Interventions: Behavioral: Supine position
- Prone Position (Experimental): It is the position where the patient lies face down with his/her head turned to the side. Arms are stretched to both sides of the head. The prone position (prone lying) is a relaxing and resting position.
  Interventions: Behavioral: Prone position
- Lateral position (Experimental): Lateral position is the left or right lateral lying position. The lateral position is given to the patient to provide proper anatomical lying and to reduce lateral flexion of the back and the strain of the large back muscles. This position prevents pressure on the bones in the back.
  Interventions: Behavioral: Lateral position

INTERVENTIONS:
Behavioral: Supine position — After the infants are treated and fed, they will be given the supine position. After positioning, the residue control will be performed in accordance with the procedure steps guideline at the 30th, 60th and 120th minutes and it will be recorded on residue follow-up form. In addition, the comfort level, heart rate, respiratory rate, and oxygen saturation levels of the infant will be evaluated and recorded at the specified times. At the end of two hours, until the next feeding hour (between 121st-180th minutes), the routine position (supine position) applied in the clinic will be given to the infant and waited in order for physiological parameters and comfort levels to return the period without intervention. The aim here is to ensure for the case to get over the effect of the previous position. No data will be collected within this period.
  Arms: Supine Position
Behavioral: Prone position — After the infants are treated and fed, they will be given the prone position. After positioning, the residue control will be performed in accordance with the procedure steps guideline at the 30th, 60th and 120th minutes and it will be recorded on residue follow-up form. In addition, the comfort level, heart rate, respiratory rate, and oxygen saturation levels of the infant will be evaluated and recorded at the specified times. At the end of two hours, until the next feeding hour (between 121st-180th minutes), the routine position (supine position) applied in the clinic will be given to the infant and waited in order for physiological parameters and comfort levels to return the period without intervention. The aim here is to ensure for the case to get over the effect of the previous position. No data will be collected within this period.
  Arms: Prone Position
Behavioral: Lateral position — After the infants are treated and fed, they will be given the left or right position. After positioning, the residue control will be performed in accordance with the procedure steps guideline at the 30th, 60th and 120th minutes and it will be recorded on residue follow-up form. In addition, the comfort level, heart rate, respiratory rate, and oxygen saturation levels of the infant will be evaluated and recorded at the specified times. At the end of two hours, until the next feeding hour (between 121st-180th minutes), the routine position (supine position) applied in the clinic will be given to the infant and waited in order for physiological parameters and comfort levels to return the period without intervention. The aim here is to ensure for the case to get over the effect of the previous position. No data will be collected within this period. These processes will continue until the 4 positions are completed. Infants will stay in each position for 2 hours.
  Arms: Lateral position

SUMMARY:
The purpose of this randomized controlled trial is to determine the effect of different positions (supine, prone, right lateral and left lateral) in post-op term newborns staying in Pediatric Cardio Vascular Surgery (PCVS) Intensive Care Unit on gastric residual volume and comfort level.

DETAILED DESCRIPTION:
In the study, crossover design from experimental designs was preferred. Crossover design is an experimental design type in which two or more interventions are applied in a sequence to each case in the study group. In these studies, each group is its own control group. In this design type, all different interventions in the study are applied to the same case; thus, differences that may arise due to individual differences are prevented. Additionally, less number of cases is sufficient in order to obtain the same number of observation data compared to the other design examples. Due to these properties, randomized crossover design model was used in this study. The study will be conducted in PCVS Intensive Care Unit of a University Hospital in Turkey between October 2020 and August 2021.

In this study, sample size was calculated at the confidence interval of 95% using "G. Power-3.1.9.4" program. In a study the effect size used for determining the sample size in the study was found to be 0.54 based on the mean and standard deviation values of the study. By using this effect size, minimum sample size was found as 38 children in order for the gastric residue amount difference between positions to express statistically significance (p<0.05) with theoretical power of 0.95. By considering that there might be losses in the study, it is planned to include a total of 44 children in the study.

The order of the 4 positions to be given to the infants in the study group (A:Prone Position, B:Right lateral Position, C:Left lateral Position, D:Supine Position) was determined by lot method. 4 different orders were chosen randomly from all possible orders of 4 positions to be given to the infants in the study group (24 different orders). Each different order of the positions was expressed as a group. 4 orders randomly selected from 24 different orders were as follows:

The order in the first group is A, C, D, and B; The order in the second group is D, A, B, and C; The order in the third group is C, B, A, and D; The order in the fourth group is B, D, C, and A.

Groups and position orders according to the result of the draw:

1. st GROUP ORDER; Prone (A), Left lateral (C), Supine (D), and Right lateral (B)
2. nd GROUP ORDER; Supine (D), Prone (A), Right lateral (B), and Left lateral (C)
3. rd GROUP ORDER; Left lateral (C), Right lateral (B), Prone (A), and Supine (D)
4. th GROUP ORDER; Right lateral (B), Supine (D), Left lateral (C), and Prone (A)

Assigning the infants to 4 groups was made in Microsoft Excel program using "RANDBETWEEN" command. All positions will be applied once to each infant. The newborns to be assigned to the groups according to this result are stated in the below table.

Groups Newborns

1. st group A, C, D, B 1, 5, 10, 11, 12, 20, 21, 30, 36, 38, 44
2. nd group D, A, B, C 19, 22, 23, 24, 25, 27, 28, 31, 32, 33, 42
3. rd group C, B, A, D 3, 4, 6, 7, 9, 13, 15, 29, 34, 37, 43
4. th group B, D, C, A 2, 8, 14, 16, 17, 18, 26, 35, 39, 40, 41

Data Collection tools:

In the data collection, "Information Form" prepared by the researcher to record the descriptive information of the newborn, "Newborn Comfort Behavior Scale" to evaluate the comfort level and "Residue Follow-up Form" to record the residual amount and the "Vital Signs Follow-up Form" to record the vital signs will be used.

Information Form: It is a form prepared by the researcher in line with the literature to record the natal and postnatal information of the newborn. The information in this form will be filled out by the researcher.

Newborn Comfort Behavior Scale: It is a Likert-type scale developed to be used to assess sedation and comfort needs, pain, and distress of newborns followed-up in the intensive care. The Newborn Comfort Behavior Scale will be evaluated at the 30th, 60th and 120th minutes after the position. The comfort level scale scoring will be evaluated and filled by the researcher and a second observer working in the Intensive Care Unit for 5 years.

Residue Follow-up Form: The form prepared to follow up the residue includes the position given, amount of nutrition, the way of feeding, feeding type, and residue amount control. The researcher will evaluate and fill out the form at the 30th, 60th and 120th minutes after feeding.

Vital Signs Follow-up Form: This form prepared by the researcher in line with the literature was composed of the parameters of heart rate (min), respiratory rate (min) and oxygen saturation value (%SpO2) of the newborn. The researcher will evaluate and fill out the form at the 30th, 60th and 120th minutes after positioning.

ELIGIBILITY:
Inclusion Criteria:

* • Having a gestational week of 37 and above,

  * Undergoing heart surgery,
  * Being separated from the mechanical ventilator,
  * Starting to be fed with nasogastric or orogastric tube,
  * Not showing any signs of infection,
  * Not using narcotic drugs in post-op period,
  * Having no factors that can interfere with feeding (vomiting, distention, necrotizing enterocolitis, etc.)
  * Having no condition that can prevent positioning,
  * Receiving Informed Consent Form from their families.

Exclusion Criteria:

* • Having a gestational week of less than 36+6 days,

  * Have not been separated from the mechanical ventilator,
  * Showing any signs of infection,
  * Using narcotic drugs in the post-op period,
  * Having factors that may prevent feeding (vomiting, distention, necrotizing enterocolitis, etc.)
  * Having a condition that can prevent positioning,
  * Receiving no consent from their mother or father.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Neonatal Comfort Behavior Scale (COMFORTneo):"change" will be assessed | The Newborn Comfort Behavior Scale will be evaluated at the 30 to 120 minutes after the position.
  This scale is a Likert type scale developed to be used in the evaluation of sedation and comfort needs, pain and distress of newborns followed-up in intensive care. COMFORTneo is composed of six parameters including alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tone. Each item in the scale is scored from 1 to 5. It is evaluated over the total score. The lowest score of COMFORTneo is 6 and the highest score is 30. If total score of the scale is between 9-13 points, it refers that the infant is "comfortable". If it is between 14-30 points, it is emphasized that the infant has "pain or distress", is uncomfortable and requires interventions that will provide comfort.
Residue Follow-up Form: "change" will be assessed | It will be checked at 30 to 120 minutes after feeding.
  The form prepared to follow up the residue includes the position given, amount of nutrition, the way of feeding, feeding type, and residue amount control.
Vital Signs Follow-up Form: "change" will be assessed | It will be evaluated at 30 to 120 minutes after positioning.
  This form prepared by the researcher in line with the literature was composed of the parameters of heart rate (min), respiratory rate (min) and oxygen saturation value (%SpO2) of the newborn.

SECONDARY OUTCOMES:
Heart Rate (min): "change" will be assessed | It will be evaluated at 30 to 120 minutes after positioning.
  The heart rate per minute will be obtained using a pulse oximeter device. A separate pulse oximeter probe will be placed on each of the infants.
Oxygen Saturation (%SpO2): "change" will be assessed | It will be evaluated at 30 to 120 minutes after positioning.
  Oxygen saturation (SpO2) will be obtained using a pulse oximeter device. A separate pulse oximeter probe will be placed on each of the infants. Pulse oximeter is a noninvasive, painless, and reliable method used to measure oxygen saturation (SpO2) in arterial blood. The rate of hemoglobin carrying oxygen in arterial blood is measured and the qualifying result is defined as functional oxygen saturation.
Respiration Rate (min): "change" will be assessed | It will be evaluated at 30 to 120 minutes after positioning.
  The respiration rate is the number of inspirations per minute. It is counted by chest movements or auscultation.

CONTACTS AND LOCATIONS:
Overall Officials: fatma yılmaz kurt, Principal Investigator — Çanakkale Onsekiz Mart University
Locations (1):
- Fatma Yılmaz Kurt, Çanakkale, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Yayan EH, Kucukoglu S, Dag YS, Karsavuran Boyraz N. Does the Post-Feeding Position Affect Gastric Residue in Preterm Infants? Breastfeed Med. 2018 Jul/Aug;13(6):438-443. doi: 10.1089/bfm.2018.0028. PMID 30016174
- [Result] Khatony A, Abdi A, Karimi B, Aghaei A, Brojeni HS. The effects of position on gastric residual volume of premature infants in NICU. Ital J Pediatr. 2019 Jan 8;45(1):6. doi: 10.1186/s13052-018-0591-9. PMID 30621733
- [Result] Ozdel D, Sari HY. Effects of the prone position and kangaroo care on gastric residual volume, vital signs and comfort in preterm infants. Jpn J Nurs Sci. 2020 Jan;17(1):e12287. doi: 10.1111/jjns.12287. Epub 2019 Oct 23. PMID 31642602
- [Result] Kaur V, Kaur R, Saini SS. Comparison of Three Nursing Positions for Reducing Gastric Residuals in Preterm Neonates: A Randomized Crossover Trial. Indian Pediatr. 2018 Jul 15;55(7):568-572. PMID 30129537
- [Result] Chen SS, Tzeng YL, Gau BS, Kuo PC, Chen JY. Effects of prone and supine positioning on gastric residuals in preterm infants: a time series with cross-over study. Int J Nurs Stud. 2013 Nov;50(11):1459-67. doi: 10.1016/j.ijnurstu.2013.02.009. Epub 2013 Mar 26. PMID 23537895